CLINICAL TRIAL: NCT01203696
Title: Effect of Amlodipine on Platelet Inhibition by Clopidogrel in Patients With Ischemic Heart Disease- a Prospective Randomized Controlled Trial
Brief Title: Effect of Amlodipine on Anti-platelet Drug Effect in Patients With Coronary Artery Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ruttonjee Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Aml-Clo-protocol-v1
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Ischemic Heart Disease
Keywords: Clopidogrel; Platelet reactivity; Amlodipine
MeSH Terms: conditions — Myocardial Ischemia | interventions — Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- non-amlodipine (Active Comparator): For patient with suboptimal angina control: anti-anginal agent excluding calcium channel blocker
  Interventions: Drug: Amlodipine
- non - amlodipine (Active Comparator): For patient with suboptimal BP control: anti-hypertensive agent excluding calcium channel blocker
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Amlodipine — For patient with suboptimal angina control: oral 2.5-10mg daily
  Other Names: Norvasc
  Arms: non-amlodipine
Drug: Amlodipine — For patient with suboptimal BP control: 2.5-10mg daily po
  Other Names: Norvasc
  Arms: non - amlodipine

SUMMARY:
Clopidogrel can reduce risk of cardiovascular disease by inhibiting platelet aggregation. It is metabolized to an active drug by a liver enzyme. Its efficacy may be measured by blood sampling for platelet activity, analyzed by VerifyNow device. Calcium Channel blocker (CCB) is also commonly used for blood pressure and anginal control in these patients. Dihydropyridine group of calcium channel blocker (e.g. amlodipine) inhibits this enzyme. There are observational studies reporting dihydropyridine CCB reducing clopidogrel effect, but the clinical implication is unclear.

This study test the hypothesis that there is no significant effect of dihydropyridines CCB on clopidogrel response compared with control. After giving consent, patients with suboptimal blood pressure or anginal control will be randomized to receive either dihydropyridine CCB or non-CCB as placebo. These patient will be follow-up in 1 month.

DETAILED DESCRIPTION:
Clopidogrel is a pro-drug, which requires hepatic transformation by the cytochrome P450 isoform 3A4 to generate the active metabolite. It inhibits adenosine-5-diphosphate (ADP)-induced platelet aggregation by irreversibly blocking the platelet P2Y12 receptor. However, response to clopidogrel shows wide individual variability, and patients with high on-treatment residual ADP-induced platelet reactivity are at an increased risk of adverse cardiovascular events. Previous study suggest co-administration of CCBs is associated with decreased platelet inhibition by clopidogrel, but these observational studies are confounded by patient's characteristics baseline difference such as proportion of hypertension and diabetes.

The objective of this randomized controlled study is to compare amlodipine with placebo on anti-platelet effect of clopidogrel.

ELIGIBILITY:
Inclusion Criteria:

* ischemic heart disease patient, and
* given loading or maintenance dose of clopidogrel and in need of it for 1 or more month
* and in need of additional drug for optimal BP control (aim blood pressure <130/90) or angina control.

Exclusion Criteria:

* existing use of amlodipine
* thrombocytopenia
* end stage renal failure
* allergy to clopidogrel/ amlodipine
* pregnancy/ lactation
* strong inhibitor or inducer of cytochrome P450 3A4 enzyme within 7 days before start of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2010-07; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Platelet reactivity unit | baseline and 4 th week
  Platelet reactivity unit as measured by VerifyNow system

SECONDARY OUTCOMES:
Percentage inhibition of platelet activity | baseline and 4th week
  Percentage inhibition of platelet activity measured by VerifyNow system

CONTACTS AND LOCATIONS:
Overall Officials: Andrew YW Li, MB, Principal Investigator — Ruttonjee Hospital
Locations (1):
- Ruttonjee Hospital, Hong Kong SAR, China

REFERENCES:
- [Derived] Li AY, Ng FH, Chan FK, Tunggal P, Chan K, Lau YK. Effect of amlodipine on platelet inhibition by clopidogrel in patients with ischaemic heart disease: a randomised, controlled trial. Heart. 2013 Apr;99(7):468-73. doi: 10.1136/heartjnl-2012-302801. Epub 2012 Oct 31. PMID 23118347